CLINICAL TRIAL: NCT02040376
Title: Placebo Controlled Double Blind Crossover Trial of Metformin for Brain Repair in Children With Cranial-Spinal Radiation for Medulloblastoma
Brief Title: Metformin for Brain Repair in Children With Cranial-Spinal Radiation for Medulloblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Donald Mabbott, Psychologist, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000039383
Record Dates: First submitted 2014-01-07; First posted 2014-01-20 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Brain Tumor Treated With Cranial or Cranial-Spinal Radiation
Keywords: Paediatrics; Medulloblastoma; Metformin
MeSH Terms: conditions — Medulloblastoma | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Crossover Group 1) (Experimental): Subjects assigned to this arm will receive metformin first, followed by a washout period and then placebo.
  Interventions: Drug: Metformin; Drug: Placebo
- Group B (Crossover Group 2) (Experimental): Subjects assigned to this arm will receive placebo first, followed by a washout period and then metformin.
  Interventions: Drug: Metformin; Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin doses will be 500 mg/m2 po daily given in 2 doses for one week and if there are no concerns increased to 1000 mg/m2 po daily given in 2 doses for the rest of the 12 week trial. The investigators will use the closest dose according to body surface area (250-500-750-1000) BID.
Drug: Placebo — Placebo doses will be 500 mg/m2 po daily given in 2 doses for one week and if there are no concerns increased to 1000 mg/m2 po daily given in 2 doses for the rest of the 12 week trial. The investigators will use the closest dose according to body surface area (250-500-750-1000) BID.

SUMMARY:
A placebo controlled double blind crossover trial of metformin in 30 children treated with radiation for medulloblastoma - the most common malignant brain tumour. The investigators used tests of thinking and learning and brain imaging techniques to examine whether metformin can enhance cognition or promote brain repair following radiation-induced brain injury.

DETAILED DESCRIPTION:
We conducted a pilot randomized, double-blind, placebo-controlled trial with crossover in survivors of pediatric brain tumors with primary endpoints of safety and feasibility and secondary endpoints of cognitive and magnetic resonance imaging (MRI) measures. Twenty-four participants were enrolled and randomly assigned to complete 12-week cycles of metformin (A) and placebo (B) in either a group AB (AB) or group BA (BA) sequence. At the point of crossover, there was a 10-week washout period in which neither group received any treatment. During the first week of each treatment cycle, a daily dose of 500 mg/m2 of metformin or placebo was administered orally. The dose was increased to 1000mg/m2 daily beginning in the second week and continuing for the remainder of the 12-week cycle.

Test procedures (Clinical & current medications reviews, Blood draws, and MRI and Cognitive testing) were performed at 4 times points during the study: 1. at study entry (Baseline 1), 2. after 12 weeks of treatment (Outcome 1), 3. after a 10-week washout period at 22 weeks (Baseline 2), and 4. At the end of the trial at 34 weeks (Outcome 2).

ELIGIBILITY:
Inclusion criteria: Survivors will be included if they:

1. Have been treated with cranial or cranial-spinal radiation,
2. Are between 5 and 21 years of age at time of consent, and
3. Either declare English as their native language or have had at least two years of schooling in English at the time of their baseline assessment.
4. Have been diagnosed with a brain tumour requiring treatment with cranial or cranial-spinal radiation at least 2 years ago, is not receiving active treatment and no more than 15 years may have elapsed between treatment with cranial-spinal radiation and time of the trial. Survivors with a shunt will be included in the trial, but will need to be identified prior to study enrollment to discuss any specific considerations for imaging.
5. Meet criteria for adequate organ function requirements:

   1. Adequate renal function defined as: Creatinine clearance or radioisotope glomerular filtration rate (GFR) > 70ml/min/1.73 m2 or serum creatinine based on age/gender as follows:

      Maximum Serum Creatinine Level (mg/dL)

      5 to < 10 years: Male = 1; Female = 1

      10 to < 13 years: Male = 1.2; Female = 1.2

      13 to < 16 years: Male = 1.5; Female = 1.4

      ≥ 16 years: Male = 1.7; Female = 1.4
   2. Adequate liver function defined as:

   Total bilirubin < 1.5 x upper limit of normal (ULN) for age, and,

   serum glutamate oxaloacetate transaminase (SGOT) (AST) or serum glutamate pyruvate transaminase (SGPT) (ALT) < 3 x upper limit of normal (ULN) for age.
6. Females of childbearing potential must have a negative pregnancy test result and must agree to use a medically acceptable method of contraception throughout the entire study period and for 30 days after the last dose of study drug.
7. Informed consent will be obtained from the participants and/or their legal guardians by study team members authorized to consent for this study.

Exclusion criteria: Survivors will be excluded if they

1. Are receiving palliative care.
2. Are unable to participate in neuro-imaging without sedation as this is the primary outcome measure for the trial.
3. Are unable to swallow tablets.
4. Are unstable and/or insulin-dependent (Type 1) diabetic patients.
5. Have acute or chronic metabolic acidosis and/or lactic acidosis.
6. Any female patient or partner who has reached menarche and male patients who are not willing to use an effective method of contraception.
7. Patient who is pregnant or lactating and does not agree to stop breastfeeding while receiving trial treatment.
8. Have a history of renal disease or renal dysfunction e.g., as suggested by elevated serum creatinine levels (see 5.a. Inclusion criteria) or abnormal creatinine clearance.
9. Have a history of congestive heart failure requiring pharmacologic treatment.
10. Have a known hypersensitivity to metformin hydrochloride.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2014-06-13 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Feasibility: Medication Adherence | Outcome 2 (Week 35)
  Participant's adherence to taking study medication (Metformin or Placebo) as instructed based on dosing nomogram, for the whole study.
  % Medication adherence = (Number of tablets actually consumed / Number of tablets expected to be consumed)*100
  Number of tablets actually consumed is based on compliance counts conducted at the end of the study.
Safety: Frequency of Adverse Events (AE) | Outcome 2 (Week 35)
  The frequency of all AEs experienced during metformin and placebo treatment for all participants.

SECONDARY OUTCOMES:
Cognitive Testing: Declarative Memory - Change in Children's Auditory Verbal Learning Test -2 (CAVLT-2) | Baseline 1 (Week 1), Outcome 1 (Week 13), Baseline 2 (Week 23), and Outcome 2 (Week 35)
  For Arm AB:
  1. Change in Immediate Recall test from Baseline 1 (Week 1) at Outcome 1 (Week 13, post 12-week intervention)
  2. Change in Immediate Recall test from Baseline 2 (Week 23, post 10-week washout) at Outcome 2 (Week 35, post 2nd 12-week intervention)
  3. Change in Immediate Recall test from Baseline 1 (Week 1) at Outcome 2 (Week 35, post 2nd 12-week intervention)
  For Arm BA:
  1. Change in Immediate Recall test from Baseline 1 (Week 1) at Outcome 1 (Week 13)
  2. Change in Immediate Recall test from Baseline 2 (Week 23) at Outcome 2 (Week 35)
  3. Change in Immediate Recall test from Baseline 1 (Week 1) at Outcome 2 (Week 35)
Cognitive Testing: Working Memory - Change in List Sort Working Memory Subtest of the NIH Toolbox Cognition Battery | Baseline 1 (Week 1), Outcome 1 (Week 13), Baseline 2 (Week 23), Outcome 2 (Week 35)
  For Arm AB:
  1. Change in List Sort Working Memory Test from Baseline 1 (Week 1) at Outcome 1 (Week 13)
  2. Change in List Sort Working Memory Test from Baseline 2 (Week 23) at Outcome 2 (Week 35)
  3. Change in List Sort Working Memory Test from Baseline 1 (Week 1) at Outcome 2 (Week 35)
  For Arm BA:
  1. Change in List Sort Working Memory Test from Baseline 1 (Week 1) at Outcome 1 (Week 13)
  2. Change in List Sort Working Memory Test from Baseline 2 (Week 23) at Outcome 2 (Week 35)
  3. Change in List Sort Working Memory Test from Baseline 1 (Week 1) at Outcome 2 (Week 35)
Cognitive Testing: Processing Speed - Change in Mean Reaction Time across Cambridge Neuropsychological Test Automated Battery (CANTAB) subtests | Baseline 1 (Week 1), Outcome 1 (Week 13), Baseline 2 (Week 23), and Outcome 2 (Week 35)
  Change in Mean Reaction Time (MRT) across the following CANTAB subtests:
  1. Rapid Visual Information Processing (RVP)
  2. Reaction Time (RT)
  3. Match to Sample Visual Search (MTS)
  4. Delayed Matching in sample (DMS)
  Each subtest provides an outcome measure of response latency, which will be averaged across all correct trials for each subtest to provide an overall measure of processing speed.
  For Arm AB:
  1. Change in MRT from Baseline 1 (Week 1) at Outcome 1 (Week 13)
  2. Change in MRT from Baseline 2 (Week 23) at Outcome 2 (Week 35)
  3. Change in MRT from Baseline 1 (Week 1) at Outcome 2 (Week 35)
  For Arm BA:
  1. Change in MRT from Baseline 1 (Week 1) at Outcome 1 (Week 13)
  2. Change in MRT from Baseline 2 (Week 23) at Outcome 2 (Week 35)
  3. Change in MRT from Baseline 1 (Week 1) at Outcome 2 (Week 35)

OTHER OUTCOMES:
Neuroimaging: MRI Measures of White Matter Growth within the Corpus Callosum | Baseline 1 (Week 1), Outcome 1 (Week 13), Baseline 2 (Week 23), and Outcome 2 (Week 35)
  Change in Axonal Water Fraction (AWF)- Diffusion Kurtosis Imaging (DKI) metric sensitive to myelin
Neuroimaging: MRI Measures of Hippocampal Volume | Baseline 1 (Week 1), Outcome 1 (Week 13), Baseline 2 (Week 23), and Outcome 2 (Week 35
  Change in Hippocampal Volume, as measured by Cerebral Blood Flow (CBF)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Mabbott, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayoub R, Ruddy RM, Cox E, Oyefiade A, Derkach D, Laughlin S, Ades-Aron B, Shirzadi Z, Fieremans E, MacIntosh BJ, de Medeiros CB, Skocic J, Bouffet E, Miller FD, Morshead CM, Mabbott DJ. Assessment of cognitive and neural recovery in survivors of pediatric brain tumors in a pilot clinical trial using metformin. Nat Med. 2020 Aug;26(8):1285-1294. doi: 10.1038/s41591-020-0985-2. Epub 2020 Jul 27. PMID 32719487